CLINICAL TRIAL: NCT06281769
Title: Clinical Validation of Transrectal Multiparametric Ultrasound Imaging Strategy (PCaVision) for the Detection of Clinically Significant Prostate Cancer: a Head-to-head Comparison With the MRI-based Strategy
Brief Title: Prostate Cancer Detection Rate of Targeted Biopsies With PCaVision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Angiogenesis Analytics (Industry)
Responsible Party: Principal Investigator, Harrie P. Beerlage, Prof.dr. H.P. Beerlage, Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL82101.000.22
Record Dates: First submitted 2024-02-12; First posted 2024-02-28 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: contrast enhanced ultrasound; CEUS; Multiparametric Ultrasound; Artificial intelligence; MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic evaluation of prostate cancer (Other)
  Interventions: Diagnostic Test: 3D multi-parametric ultrasound targeted biopsy pathway using PcaVision; Diagnostic Test: MRI targeted biopsy pathway

INTERVENTIONS:
Diagnostic Test: 3D multi-parametric ultrasound targeted biopsy pathway using PcaVision — The procedure of 3D multiparametric ultrasound consists of 3 components: (1) intravenous administration of ultrasound contrast; (2) rectal multi-parametric ultrasound imaging; (3) PCaVision: artificial intelligence algorithm analyzing the images.
Diagnostic Test: MRI targeted biopsy pathway — MRI sequences will include at least T1-weighted, T2-weighted, Diffusion-weighted imaging (DWI) and calculation of apparent diffusion coefficient (ADC) maps. Scoring of suspicion will be performed using the European Society of Urogenital Radiology (ESUR) PI-RADS standardized scoring system. All lesions will be marked and delineated for MRI-TRUS fusion 3D multiparametric ultrasound (mpUS).

SUMMARY:
The primary objective is to demonstrate non-inferiority of the detection rate of clinically significant prostate cancer (csPCa) in targeted biopsies based on PCaVision imaging (PCaVision pathway) in comparison with the detection rate of clinically significant cancer in targeted biopsies based on MRI (MRI pathway).

DETAILED DESCRIPTION:
All patients will undergo imaging using MRI and PCaVision during which suspicious lesions will be identified based on each imaging technique independently with readers being blinded for the results of the other imaging technique. Thereafter, a MRI targeted 3-core biopsy per lesion (maximum of 2 lesions) and/ or a PCaVision targeted 3-core biopsy (maximum of 2 lesions) will be performed by a one physician if suspicious lesions have been identified based on imaging. If lesions have been identified with both PCaVision and MRI in the same patient, the order of the targeted biopsies will be randomized. If the same lesion has been identified on both MRI and PCaVision, both a MRI-targeted and a PCaVision targeted biopsy will be separately performed. Histological examination of the targeted biopsies will be performed to determine presence of clinically significant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* be male
* have an age of 18 years or older
* be biopsy naïve
* have a clinical suspicion of prostate cancer
* be scheduled for evaluation by prostate MRI based on a suspicious DRE and/or elevated serum PSA
* have signed informed consent

Exclusion Criteria:

* active (urinary tract) infection or prostatitis
* a patient history with a cardiac right-to-left shunt.
* allergic to sulphur hexafluoride or any of the other ingredients of the ultrasound contrast agent SonoVue
* current treatment with dobutamine
* known severe pulmonary hypertension (pulmonary artery pressure >90 mmHg), uncontrolled systemic hypertension or respiratory distress syndrome
* any (further) contraindication to undergo MRI or 3D mpUS imaging
* incapable of understanding the language in which the patient information is given.
* medical history of prostate surgery
* treatment of 5 alpha-reductase inhibitors for at least 3 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Detection rate of clinically significant prostate cancer (csPCa) in targeted biopsies based on PCaVision imaging in comparison with the detection rate of clinically significant cancer in targeted biopsies based on MRI. | Two weeks
  csPCa defined as GG ≥ 2 in any of the biopsy cores taken from a lesion

SECONDARY OUTCOMES:
Proportion of men in whom targeted biopsies could be safely omitted in the PCaVision pathway versus the MRI pathway. | Two weeks
  Defined as the number of men in whom no lesions for target biopsies have been identified by PCaVision while no CsPCa is detected in either MRI targeted biopsies or systematic biopsies.
Detection rate of three different definitions of prostate cancer in targeted biopsies based on PCaVision imaging (PCaVision pathway) in comparison with the detection rate of targeted biopsies based on MRI (MRI pathway). | Two weeks
  (i) ISUP ≥ 3 in any of the biopsy cores taken from a lesion; (ii) ISUP ≥ 2 with cribriform growth and/or intraductal carcinoma (CR/IDC) in any of the biopsy cores taken from a lesion; (iii) ISUP = 1
Number of men in whom the PCaVision pathway generated insufficient quality images with the number of men with insufficient quality MRI images in the MRI pathway. | Two weeks
Detection rate of clinically significant prostate cancer in targeted biopsies based on PCaVision imaging using various incremental levels of PCaVision's image quality requirements in comparison with the detection rate of targeted biopsies based on MRI. | Two weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - Amsterdam UMC - location VUmc, Amsterdam
  - Andros Clinics, Baarn
  - Spaarne Gasthuis, Hoofddorp
  - St. Antonius, Nieuwegein
  - Fransiscus Gasthuis, Rotterdam

REFERENCES:
- [Background] van Moorselaar RJ, Voest EE. Angiogenesis in prostate cancer: its role in disease progression and possible therapeutic approaches. Mol Cell Endocrinol. 2002 Nov 29;197(1-2):239-50. doi: 10.1016/s0303-7207(02)00262-9. PMID 12431818
- [Background] van den Kroonenberg DL, Jager A, Garrido-Utrilla A, Reitsma JB, Postema AW, Beerlage HP, Oddens JR. Clinical Validation of Multiparametric Ultrasound for Detecting Clinically Significant Prostate Cancer Using Computer-Aided Diagnosis: A Direct Comparison with the Magnetic Resonance Imaging Pathway. Eur Urol Open Sci. 2024 Jul 1;66:60-66. doi: 10.1016/j.euros.2024.06.012. eCollection 2024 Aug. PMID 39050912
- [Result] Russo G, Mischi M, Scheepens W, De la Rosette JJ, Wijkstra H. Angiogenesis in prostate cancer: onset, progression and imaging. BJU Int. 2012 Dec;110(11 Pt C):E794-808. doi: 10.1111/j.1464-410X.2012.11444.x. Epub 2012 Sep 7. PMID 22958524
- [Result] Mischi M, Kuenen MP, Wijkstra H. Angiogenesis imaging by spatiotemporal analysis of ultrasound contrast agent dispersion kinetics. IEEE Trans Ultrason Ferroelectr Freq Control. 2012 Apr;59(4):621-9. doi: 10.1109/TUFFC.2012.2241. PMID 22547274
- [Result] Kuenen MP, Saidov TA, Wijkstra H, de la Rosette JJ, Mischi M. Spatiotemporal correlation of ultrasound contrast agent dilution curves for angiogenesis localization by dispersion imaging. IEEE Trans Ultrason Ferroelectr Freq Control. 2013 Dec;60(12):2665-9. doi: 10.1109/TUFFC.2013.2865. PMID 24297031
- [Result] Postema AW, Frinking PJ, Smeenge M, De Reijke TM, De la Rosette JJ, Tranquart F, Wijkstra H. Dynamic contrast-enhanced ultrasound parametric imaging for the detection of prostate cancer. BJU Int. 2016 Apr;117(4):598-603. doi: 10.1111/bju.13116. Epub 2015 Jun 29. PMID 25754526
- [Result] Postema AW, Gayet MCW, van Sloun RJG, Wildeboer RR, Mannaerts CK, Savci-Heijink CD, Schalk SG, Kajtazovic A, van der Poel H, Mulders PFA, Beerlage HP, Mischi M, Wijkstra H. Contrast-enhanced ultrasound with dispersion analysis for the localization of prostate cancer: correlation with radical prostatectomy specimens. World J Urol. 2020 Nov;38(11):2811-2818. doi: 10.1007/s00345-020-03103-4. Epub 2020 Feb 20. PMID 32078707
- [Result] Mannaerts CK, Engelbrecht MRW, Postema AW, van Kollenburg RAA, Hoeks CMA, Savci-Heijink CD, Van Sloun RJG, Wildeboer RR, De Reijke TM, Mischi M, Wijkstra H. Detection of clinically significant prostate cancer in biopsy-naive men: direct comparison of systematic biopsy, multiparametric MRI- and contrast-ultrasound-dispersion imaging-targeted biopsy. BJU Int. 2020 Oct;126(4):481-493. doi: 10.1111/bju.15093. Epub 2020 May 13. PMID 32315112
- [Result] Mannaerts CK, Wildeboer RR, Remmers S, van Kollenburg RAA, Kajtazovic A, Hagemann J, Postema AW, van Sloun RJG, J Roobol M, Tilki D, Mischi M, Wijkstra H, Salomon G. Multiparametric Ultrasound for Prostate Cancer Detection and Localization: Correlation of B-mode, Shear Wave Elastography and Contrast Enhanced Ultrasound with Radical Prostatectomy Specimens. J Urol. 2019 Dec;202(6):1166-1173. doi: 10.1097/JU.0000000000000415. Epub 2019 Jun 27. PMID 31246546
- [Result] Jager A, Vilanova JC, Michi M, Wijkstra H, Oddens JR. The challenge of prostate biopsy guidance in the era of mpMRI detected lesion: ultrasound-guided versus in-bore biopsy. Br J Radiol. 2022 Mar 1;95(1131):20210363. doi: 10.1259/bjr.20210363. Epub 2021 Jul 29. PMID 34324383
- See also: Clinical Trial Protocol: Developing an Image Classification Algorithm for Prostate Cancer Diagnosis on Three-dimensional Multiparametric Transrectal Ultrasound — https://doi.org/10.1016/j.euros.2022.12.018

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT06281769/Prot_SAP_002.pdf